CLINICAL TRIAL: NCT04402996
Title: Evaluation of Meteorin-like Levels in Individuals With Healthy and Periodontal Disease
Brief Title: Meteorin-like Levels in Individuals With Periodontitis
Status: Completed | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Ebru SAĞLAM, Principal Investigator,Health Sciences University, Dentistry Faculty, Istanbul Saglik Bilimleri University
Other Study IDs: Sağlık Bilimleri Üniversitesi
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Periodontitis; Gingivitis; Healthy
Keywords: Meteorin-like
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Gingival Crevicular Fluid and Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Individuals with Periodontally Healthy
  Interventions: Other: Saliva; Other: gingival crevicular fluid
- Gingivitis: Individuals with Gingival Inflammation
  Interventions: Other: Saliva; Other: gingival crevicular fluid
- Periodontitis: Individuals with Periodontitis
  Interventions: Other: Saliva; Other: gingival crevicular fluid

INTERVENTIONS:
Other: Saliva — individuals' saliva samples will be collected and transferred to eppendorf tubes.
  Until biochemical analysis is carried out will be stored in -80ºC.
  Other Names: sampling
Other: gingival crevicular fluid — GCF samples of individuals will be collected by paper strips and transferred to eppendorf tubes.
  Until biochemical analysis is carried out will be stored in -80ºC.
  Other Names: sampling

SUMMARY:
Metrnl has proven to be an inflammatory-related immunoregulatory cytokine and shown to play a role in the pathogenesis of human inflammatory diseases. Metrnl is highly expressed from the oral mucosa to the esophagus. Periodontitis is a chronic inflammatory disease that can start with localized inflammatory reactions created by the supporting tissues surrounding the teeth against microorganisms and then result in loss of teeth. The authors think that Metrnl may play a role in the periodontitis. The aim of this study is to compare the Metrnl, IL-1β, and IL-10 levels of healthy and periodontitis individuals.

DETAILED DESCRIPTION:
Periodontitis is a destructive chronic inflammatory disease that can start with localized inflammatory reactions created by the supporting tissues surrounding the teeth against microorganisms and then result in loss of teeth. Cytokines play an important role in inflammation that occurs in periodontal disease.

Interleukine -1β ( IL-1β ) levels are associated with periodontal destruction in the pathogenesis of periodontal disease. Cytokines such as Interleukine-10 (IL-10) and transforming growth factor- β (TGF-β) have been reported to decrease periodontal disease progression rate.

Gingival crevicular fluid shows the cellular response in the periodontium. The most important host-related ingredients are inflammatory markers, including cytokines, enzymes, and interleukins. Saliva analysis is used in the diagnosis of systemic conditions as well as in the diagnosis of oral pathologies.

Meteorin- like (Metrnl) is a protein that plays a role in natural and acquired immune-related functions and inflammatory responses, and expressed in barrier tissues (skin and mucosa) as well as various macrophage populations, from dendritic cells and some granulocytes. Metrnl has proven to be an inflammatory-related immunoregulatory cytokine and shown to play a role in the pathogenesis of human inflammatory diseases. Metrnl, which is highly expressed from the oral mucosa to the esophagus, may play a role in the onset of periodontitis and an effective marker in preventing the progression of destruction. We think that Metrnl plays an important role in periodontitis, an inflammatory disease. The aim of this study is to compare the Metrnl, IL-1β, and IL-10 levels of healthy and periodontitis individuals

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* individuals who does not have a disease under treatment,
* individuals without regular systemic medication

Exclusion Criteria:

* smoking
* receiving periodontal treatment in the last 6 months
* pregnancy
* menopausal or menstrual period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals will be divided into three different groups, about 20-25 people in each group.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
IL-1β | through study completion, an average of 6 months
  saliva and serum levels
Metrnl | through study completion, an average of 6 months
  saliva and serum levels
IL-10 levels | through study completion, an average of 6 months
  saliva and serum levels

SECONDARY OUTCOMES:
Plaque Index | up to 20 weeks
  Silness-Löe
Probing Depth | up to 20 weeks
  millimeter
Bleeding on Probe | up to 20 weeks
  Ainamo&Bay

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Toraman, Dr., Study Chair — Saglik Bilimleri Universitesi; Serhat Köseoğlu, assoc prof, Study Chair — Saglik Bilimleri Universitesi; Mehmet Sağlam, assoc prof, Study Chair — Izmir Katip Celebi University; Levent Savran, PhD, Study Chair — Izmir Katip Celebi University; Ebru Sağlam, Dr, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Ebru Sağlam, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No